CLINICAL TRIAL: NCT03664492
Title: Talking About Weight With Families: An Innovative Educational Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Staff endocrinologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000055748
Record Dates: First submitted 2018-02-01; First posted 2018-09-10 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Childhood Obesity
Keywords: Communication about weight; education; parents; health care professionals
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: The recruited group of health care professionals/parents will answer a pre-questionnaire, then watch an educational video, then answer a post-questionnaire. If they agree, these participants will be asked to complete a third questionnaire (retention questionnaire) 4 to 6 months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Whiteboard video (Other): All the interested participants contacting us will be provided an info email and an internet link via email to access the study through REDCap. Participants will be prompted to complete pre-questionnaire, followed by access to the video, with a prompt to complete the post questionnaire after. If they agree, they will receive 4 to 6 months later, a third questionnaire to complete. For those without access to the internet, we will offer to them view the video at the SickKids at their convenience.
  Interventions: Other: Educational whiteboard video

INTERVENTIONS:
Other: Educational whiteboard video — Participants will be prompted to complete pre-questionnaire, followed by access to the video, with a prompt to complete the post questionnaire after. If they agree, they will receive 4 to 6 months later, a third questionnaire to complete. For those without access to the internet, we will offer to them view the video at the SickKids at their convenience.

SUMMARY:
Tools are limited to help health care professionals and parents talk about weight-related issues with their paediatric patients and children, respectively. The investigators have developed two whiteboard videos: 1) to aim to help health care professionals talk about weight-related issues with paediatric patients and their families, and 2) to aim to help parents feel more comfortable talking about weight with their children. This study aims to evaluate the videos using pre and post questionnaires. With the questionnaires, the investigators want to evaluate the content, the quality, the usability of the video and to measure how helpful the video were for health care professionals and parents.

DETAILED DESCRIPTION:
Nearly one third of Canadian children and adolescents are overweight or obese. Eating disorders are the third most common chronic condition in adolescents. Although both of these issues are highly prevalent, parents who have children struggling with either underweight or overweight are concerned about how to approach those topics. Even though they are usually well-intended, their intervention may have a negative impact. Indeed, research has shown that parents who encourage their children to diet or discuss their own diet is associated with overweight or eating disorders in their children. Conversely, if parents focus on healthful eating behaviors, overweight adolescents are less likely to diet and to use unhealthy weight-control behaviors. In that context, in order to help children struggling with unhealthy lifestyle behaviours, the development of educational materials to promote healthy and helpful conversation about weight for parents is critically needed. While the use of educational videos with parents has been studied, this will be the first study examining videos to educate parents regarding weight-related communication.

Available literature also suggests that health care professionals feel ill-equipped to address weight-related issues with their patients, particularly obesity. A lack of self-efficacy and training are recognized as two significant barriers to discussing weight with patients and their families. Other challenges include the fear of damaging their relationship with patients and their families and the apprehension of triggering other issues such as eating disorders. Thus, educational materials to help health care professionals talk about weight-related issues with their patients are warranted. Educational videos have been shown to be an effective way to improve knowledge, confidence, and attitudes of health care professionals and trainees.

The investigators have designed two whiteboard videos based on a weight-related communication scoping review and on the key messages identified in a focus groups conducted previously by our group (McPherson A et al. Talking with children and families about obesity and weight related topics: A scoping review of best practices. Obes Rev.). They will evaluate the videos using pre and post questionnaires directed on usability, content, quality (acceptability, engagement) and measuring the impact on perceived self-efficacy in regards to discussing weight. The investigators will also evaluate the impact of the video over time with a third questionnaire 4 to 6 months later. The pre questionnaire for parents will include socio-demographic questions to enable us to provide sample characteristics. These data will be collected as they are known to have impact on the way weight is perceived. The investigators hypothesize that health care professionals' perceived self-efficacy on discussing weight-related issues with their paediatric patients and parents' perceived self-efficacy on raising weight issues with their children and answering their answers on that topic will improve after watching the videos, and will persist over time.

ELIGIBILITY:
Inclusion Criteria:

* Health care professionals and trainees
* Parents with a child under 18 years old

Exclusion Criteria:

* Inability to speak and read English fluently
* Moderate to severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Post Questionnaire - Parents (4-6 mo) - Confidence in ability to raise the issue about weight | 4 - 6 months post education video
  Change in confidence level in their ability to raise the issue/talk about weight with their children using a scale from 0-100.
Post Questionnaire - Parents (4-6 mo) - Level of agreement in statements related to behvaiour change | 4 - 6 months post education video
  Level of agreement in statements related to behaviour change post education using in a 5 point likert scale
Health Care Professional Post Questionnaire - Confidence in initiating conversation about overweight | immediately post education video
  Change in confidence level for initiating a conversation with a family or pediatric patient that meets criteria for overweight or obesity using a scale from 0-100.
Health Care Professional Post Questionnaire - Confidence in initiating conversation about underweight | immediately post education video
  Change in confidence level for initiating a conversation with a family or pediatric patient that meets criteria for underweight using a scale from 0-100.
Health Care Professional Questionnaire (4-6 Months Post) Confidence in initiating conversation about overweight | 4 - 6 months post education video
  Change in confidence level for initiating a conversation with a family or pediatric patient that meets criteria for underweight using a scale from 0-100.
Health Care Professional Questionnaire (4-6 Months Post) Confidence in initiating conversation about underweight | 4 - 6 months post education video
  Change in confidence level for initiating a conversation with a family or pediatric patient that meets criteria for overweight or obesity using a scale from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Jill K Hamilton, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The investigators plan to publish in a peer reviewed journal, as well as present at national and international conferences (Canadian Pediatric Endocrine Group, International Conference for Obesity and Canadian Pediatric Society )

REFERENCES:
- [Result] Klupt KA, Oreskovich SM, Bernard-Genest J, Patel BP, Chu L, Dettmer E, Walsh CM, Strom M, McPherson AC, Strub J, Steinberg A, Steinegger C, Hamilton JK. Careful conversations: an educational video to support parents in communicating about weight with their children. BMC Pediatr. 2020 Aug 24;20(1):397. doi: 10.1186/s12887-020-02284-6. PMID 32838762
- [Derived] Bernard-Genest J, Chu L, Dettmer E, Walsh CM, McPherson AC, Strub J, Steinberg A, Steinegger C, Hamilton JK. Talking About Weight With Families-Helping Health Care Professionals Start the Conversation: A Nonrandomized Controlled Trial. Clin Pediatr (Phila). 2020 Sep;59(9-10):910-917. doi: 10.1177/0009922820922844. Epub 2020 May 30. PMID 32475155